CLINICAL TRIAL: NCT04555382
Title: Association Between CAF, L-FABP and NGAL and the Occurence of Acute Kidney Injury : a Potential Diagnostic Model of Three Biomarkers.
Brief Title: Combining CAF, L-FABP and NGAL as a Potentially Diagnostic Model for Acute Kidney Injury.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-791
Record Dates: First submitted 2020-09-15; First posted 2020-09-18 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-09

CONDITIONS: Acute Kidney Injury
Keywords: L-FABP, Acute Kidney Injury, diagnosis, biomarker
MeSH Terms: conditions — Acute Kidney Injury; Disease | interventions — Blood Specimen Collection; Urination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood and urine samples were collected from the patients every twelve hours, and time was limited with a maximum of seven days for every patients. After centrifuging with 3000rpm for 5minutes, 1.5mL of supernate was taken into EP tube and stored in the refrigerator at -80℃
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- AKI group: this group are included patients who have not occured acute kidney injury at first, however acute kidney injury are occured soon afterwards during the observation period.
  Interventions: Diagnostic Test: Blood and Urine
- non-AKI group: this group are included patients who have not occured acute kidney injury during the observation period.
  Interventions: Diagnostic Test: Blood and Urine

INTERVENTIONS:
Diagnostic Test: Blood and Urine — Blood and urine samples are collected every twelve hours when the patients are included in the study during observation period.

SUMMARY:
Acute kidney injury was a common clinical complication, and many diseases were associated with a high risk of occurrence of AKI. We explored the clinical utility of serum CAF, L-FABP and NGAL by constructing a diagnostic model for identification of ICU patients at risk for AKI and distinguish different etiologies of AKI.

This observational cohort study included one hundred patients who had been in ICU from the Second Affiliated Hospital of Zhejiang University School of Medicine between August 2020 and August 2022. Blood and urine samples were collected every 12 hours until 7 days. The time of staying with ICU less than 2 days were removed. CAF, L-FABP and NGAL was measured based on the platform of Chemiluminescent Immunoassay, and assessed the diagnostic value of the occurrence of AKI. By constructing an effective diagnostic model to provide effective clinical decision-marking for early intervention.

DETAILED DESCRIPTION:
The observational cohort study included one hundred patients who were from the intensive care unit of the Second Affiliated Hospital of Zhejiang University School of Medicine between August 2020 and August 2022. AKI was defined according to the Kidney Disease Improving Global Outcomes (KDIGO) guidelines as renal function was suddenly decreased within 48 hours and serum creatinine increased at least 0.3mg/dL, or serum creatinine increased more than 1.5 times higher than baseline within 7 days, or urine volume less than 0.5mL/Kg per hour for 6 hours. The staging criteria of AKI as follows: stage I means serum creatinine higher than baseline between 1.5times and 1.9 times, or serum creatinine increased at least 26.5μmol/L, or serum creatinine increased more than 1.5 times higher than baseline within 7 days, or urine volume less than 0.5mL/Kg per hour for 6 hours; stage II means serum creatinine higher than baseline between 2.0 times and 2.9 times, or urine volume less than 0.5mL/Kg per hour for 12hours; stage III means serum creatinine higher than baseline 3.0 times, or serum creatinine higher than baseline 353.6μmol/L, or started renal replacement therapy. Patients who stayed in the ICU for less than 24 hours and whose serum creatinine had increased above normal reference range on the first day of ICU were excluded.

Collecting the blood and urine samples of the patients regularly every twelve hours, centrifuging samples in 3000rpm for 5 minutes, freezing at -80℃, all patients' clinical information should be recorded by name, age ,sex, BMI index, hypertension, diabetes, cardiac disease, and so on. All patients have written informed contents and this study was approved by the Second Affiliated Hospital of Zhejiang University School of Medicine.NGAL, CAF and L-FABP was measured by chemiluminescent immunoassay with Robust i1000.

ELIGIBILITY:
Inclusion Criteria:

1. the serum creatinine was increased above reference range at first when patients were included intensive care unit;
2. renal dialysis and plasma exchange were never occured when patients were included in the study;
3. patients who were included in the study stayed at two days in ICU.

Exclusion Criteria:

1. patients who stayed in ICU for less than 24 hours;
2. the serum creatinine was increased above reference range before ICU admission;
3. kidney-related diseases were existed before ICU admission.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The objects of study are the patients from the intensive care unit of the Second Affiliated Hospital of Zhejiang University School of Medicine between August 2020 and August 2022.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-08-15 (Actual); Primary Completion 2022-02-15 (Estimated); Study Completion 2022-08-15 (Estimated)

PRIMARY OUTCOMES:
the concentration of CAF, L-FABP and NGAL | seven days after admission
  the concentration of CAF, L-FABP and NGAL of blood and urine samples of every patients are measured by Chemiluminescent Immunoassay

CONTACTS AND LOCATIONS:
Overall Officials: Tao Zhihua, Study Chair — 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No